CLINICAL TRIAL: NCT04413643
Title: Noninvasive Ventilation for Chronic Obstructive Pulmonary Disease: Hospital to Home Pilot
Brief Title: NIV for COPD: Hospital to Home
Acronym: H2H
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: ResMed (Industry)
Responsible Party: Principal Investigator, Kathleen Sarmiento, Staff Physician, Medicine Service, San Francisco Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-25750
Record Dates: First submitted 2019-10-07; First posted 2020-06-04 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Noninvasive Ventilation
Keywords: COPD; BIPAP; NIV; Respiratory failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: This is a feasibility trial intended to inform a larger clinical trial based on outcomes data collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Noninvasive Ventilation (Experimental): Subjects will be introduced to NIV and educated on sleep disordered breathing. NIV will be initiated during hospitalization following resolution of acute respiratory failure. NIV settings will be based on inspiratory and expiratory positive airway pressures (IPAP, EPAP), rates, and tidal volumes tolerated during the acute phase of treatment. Initial settings will be set with goals of tolerance and acceptance of therapy. Minimum pressure difference between IPAP and EPAP settings will be 5cmH20. Volume assured pressure support mode with a target tidal volume (Vt) of 8ml/kg ideal body weight will be used. Final device settings and patient parameters will be documented after 10 minutes of acclimation to the device. Data from the device will be reviewed the following day. Tolerance, mask comfort, and acceptance of therapy will be assessed. Changes to settings, mask interface, or other comfort features will be performed at this initial reassessment period.
  Interventions: Device: Noninvasive Ventilation

INTERVENTIONS:
Device: Noninvasive Ventilation — The use of non-invasive ventilation (NIV) has been extensively evaluated in both patients with stable disease in the home setting and in AECOPD during hospitalization. It is widely accepted that NIV used during AECOPD in the inpatient setting reduces rates of endotracheal intubation, as well as length of ICU and hospital stay. Long-term use of NIV, particularly at higher pressures, in the home setting in COPD patients with evidence of chronic compensated respiratory acidosis (PaCO2 >45mmHg) decreases elevated PaCo2 and serum bicarbonate levels, improves pulmonary function, and improves quality of life. Little is known about whether patients initiated on NIV during an AECOPD and subsequently transitioned to long-term home NIV on discharge demonstrate reduced AECOPD rates, readmission rates, or differences in morbidity and mortality.

SUMMARY:
This is a pilot study to evaluate the impact of providing patients admitted with acute exacerbations of COPD (AECOPD) with non-invasive ventilation (NIV)home devices prior to discharge on hospital readmission rates and other secondary outcomes.

Aim 1 To test whether continuation of NIV at home after being initiated during hospitalization for AECOPD improves subsequent admission-free survival in patients with chronic hypercapnic respiratory failure secondary to COPD

Hypothesis 1: The use of targeted NIV during hospitalization with continuation upon discharge to home will improve one-year all-cause mortality as compared to published mortality in the current literature.

Hypothesis 2: The use of targeted NIV during hospitalization with continuation upon discharge to home will reduce readmission rates for AECOPD within-institution historical data.

Aim 2 To evaluate the feasibility of a larger multisite randomized controlled trial in veterans using inclusion and exclusion criteria specified in this pilot.

Outcomes

Primary: Event-free survival (re-hospitalization for AECOPD, time to readmission for AECOPD, and all-cause mortality)

Secondary:

1. Unplanned readmission rates (all complications)
2. Time to readmissions for admissions other than AECOPD.
3. Arterial blood gas/Venous blood gas (ABG/VBG): PaO2, PaCO2 and serum bicarbonate at Baseline, 6 and 12 months
4. Pulmonary function (handheld spirometer or in-laboratory based on specific institution resources) at Baseline, 6, and 12 months 5.6 minute walk test at Baseline, 6,and 12 months

6.Health related quality of life (HRQOL) measured by the St. Georges respiratory questionnaires (SGRQ) at Baseline, 1,3,6,9 and 12 months 7.Adherence to NIV at Week 1-2, Months 1,3,6,9 and 12 8.Sleep assessed by type 3 portable monitors 9.Sleep assessed by questionnaires: Insomnia severity index (ISI), Epworth Sleepiness Scale (ESS), Pittsburgh Sleep Quality Index (PSQI), Functional Outcomes of Sleep Short Form (FOSQ-10) at Baseline, 1,3,6,9 and 12 months 11.Utilization of healthcare services (number of visits to outpatient clinics and emergency services, number of inpatient admissions)

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a leading cause of morbidity and mortality worldwide, with the economic and social burden of disease anticipated to increase annually. Acute exacerbations of COPD (AECOPD) are associated with significant in-hospital mortality (6-8%), high readmission rates (60-80%), and even more dramatic 1-year mortality (23-49%).

The use of non-invasive ventilation (NIV) has been extensively evaluated in both patients with stable disease in the home setting and in AECOPD during hospitalization. It is widely accepted that NIV used during AECOPD in the inpatient setting reduces rates of endotracheal intubation, as well as length of ICU and hospital stay. Long-term use of NIV, particularly at higher pressures, in the home setting in COPD patients with evidence of chronic compensated respiratory acidosis (PaCO2 >45mmHg) decreases elevated PaCo2 and serum bicarbonate levels, improves pulmonary function, and improves quality of life. Little is known about whether patients initiated on NIV during an AECOPD and subsequently transitioned to long-term home NIV on discharge demonstrate reduced AECOPD rates, readmission rates, or differences in morbidity and mortality. The few existing randomized trials aimed at this patient population suffer from criticisms of lack of power, varying degrees of patient symptoms, conflicting results, and inconsistent approaches in NIV strategies. Nonetheless, this is an important population to address, as AECOPD frequently leads to accelerated loss of lung function (pre-AECOPD function not recovered), decreased quality of life (QOL), more frequent exacerbations, and higher overall mortality. If NIV can minimize the loss of lung function during the transition period following AECOPD, QOL, physical activity tolerance, readmission rates and overall mortality may improve.

Economic analyses of the use of NIV in patients with AECOPD transitioning from the inpatient to home setting are also sparse, but of high value as healthcare transitions toward bundled payments and penalties for readmissions. This pilot study seeks to better inform the literature on the role of NIV initiated during inpatient AECOPD and continued long-term following discharge home in patients with chronic hypercapnic respiratory failure due to COPD. The investigators hypothesize that the use of NIV during acute inpatient treatment of AECOPD followed by continuation of NIV therapy long-term at home will improve admission free survival, improve quality of life, reduce 1-year exacerbation rates, and reduce 30d readmissions.

This is a prospective 1-year interventional pilot study that will occur at 4 Veterans Affairs (VA) hospitals (Sacramento, Durham, Pittsburgh, and San Francisco).

The total enrollment goal across all sites is 50. Total study period expected includes an enrollment period of approximately 10-12 months and follow-up period of 12 months for a total study duration of approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Admission for acute hypercapnic respiratory failure requiring mechanical ventilation or NIV
2. Resolution of acute respiratory failure reflected by normalization of pH and downgrade of clinical status to ward or floor status.
3. Severe COPD defined by GOLD stage 3 (FEV1 30-50%) or 4 (FEV1 < 30%) OR GOLD C or D. Pulmonary function tests (PFTs) done within 3 years preceding admission are acceptable to document an obstructive ventilatory defect and decrease diffusion capacity consistent with emphysema and COPD. If no PFTs are available, bedside spirometry will be performed to confirm COPD.
4. Chronic compensated respiratory acidosis based on PaCO2 >52 adjusted for pH 7.40, on pre-admission laboratory values or after resolution of acute respiratory failure.
5. Able to consent without surrogate and complete all required study visits.

Exclusion Criteria:

1. Moderate or severe obstructive sleep apnea (OSA), apnea-hypopnea index (AHI) >15/h. Sleep testing done within the prior 3 years with no increase in body mass index (BMI) >2kg/m2 or major change in cardiopulmonary conditions (new reduced ejection heart failure [HFrEF], atrial fibrillation [AFib], opioid use with morphine dose equivalent (MDDE) >120mg, or cardiothoracic surgery for lung resection or coronary artery bypass grafting) will be accepted for AHI severity.
2. BMI>35 kg/m2
3. Congestive heart failure (HFrEF, EF< 45%)
4. Other cause of chronic respiratory failure: Obesity hypoventilation syndrome, spinal cord injury (cervical or thoracic) neuromuscular disease, diaphragmatic paralysis, chest wall restrictive ventilatory defect
5. Lack of stable housing, homelessness, or unreliable electricity source in home environment.
6. Use of NIV at home within past three months
7. Failure to tolerate NIV during initial hospitalization
8. Unable or unwilling to comply with the protocol
9. Age <18 years
10. Inability to consent due to limited cognitive capacity
11. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Event-free survival | 1 year
  Re-hospitalization for AECOPD, time to readmission for AECOPD, and all-cause mortality

SECONDARY OUTCOMES:
Unplanned readmission rates (all complications) | 1 year
Time to readmissions for admissions other than AECOPD | 1 year
Change in PaO2 levels from baseline to 12mo | 1 year
  PaO2 will be measured at baseline, 6 and 12 months and evaluated for significant increase (PaO2) or decrease (PaCO2, serum bicarbonate)
Change PaCO2 levels from baseline to 12mo | 1 year
  PaCO2 will be measured at baseline, 6 and 12 months and evaluated for significant increase (PaO2) or decrease (PaCO2, serum bicarbonate)
Change in serum bicarbonate levels from baseline to 12mo | 1 year
  Serum bicarbonate will be measured at baseline, 6 and 12 months and evaluated for significant increase (PaO2) or decrease (PaCO2, serum bicarbonate)
Spirometry/Lung Function | 1 year
  Forced expiratory volume (FEV1) measured at baseline, 6mo and 12mo
Spirometry/Lung Function | 1 year
  Absolute Forced Expiratory Volume (L) measured at baseline, 6mo and 12mo
Spirometry/Lung Function | 1 year
  % Forced Expiratory Volume measured at baseline, 6mo and 12mo
Spirometry/Lung Function | 1 year
  Forced Vital Capacity (FVC) measured at baseline, 6mo and 12mo
Spirometry/Lung Function | 1 year
  Absolute Forced Vital Capacity (L) measured at baseline, 6mo and 12mo
Spirometry/Lung Function | 1 year
  % Forced Vital Capacity measured at baseline, 6mo and 12mo
Spirometry/Lung Function | 1 year
  Total Lung Capacity (TLC) measured at baseline, 6mo and 12mo
Spirometry/Lung Function | 1 year
  Absolute Total Lung Capacity (L) measured at baseline, 6mo and 12mo
Spirometry/Lung Function | 1 year
  % Total Lung Capacity measured at baseline, 6mo and 12mo
Spirometry/Lung Function | 1 year
  Residual Volume (RV) measured at baseline, 6mo and 12mo
Spirometry/Lung Function | 1 year
  Absolute Residual Volume (L) measured at baseline, 6mo and 12mo
Spirometry/Lung Function | 1 year
  % Residual Volume measured at baseline, 6mo and 12mo
Spirometry/Lung Function | 1 year
  FEV1/FVC% measured at baseline, 6mo and 12mo
Spirometry/Lung Function | 1 year
  Diffusion Capacity (DLCO) measured at baseline, 6mo and 12mo
6 minute walk test | 1 year
  At baseline, 6 mo and 12 mo
St. Georges Respiratory Questionnaire | 1 year
  50-item, 3 component questionnaire. Scores range from 0-100 with a higher score indicating more limitations. Measures the impact of breathing symptoms on quality of life. Administered at baseline, 1, 3, 6, 9 and 12 months
Adherence/Compliance with NIV | 1 year
  Standard total days used since therapy initiation (day 0). Measured at week 1-2, months 1, 3, 6, 9 and 12. Data will be obtained through remote review of wireless data transmitted from each device.
Adherence/Compliance with NIV | 1 year
  Percent days with use >4h/d. Measured at week 1-2, months 1, 3, 6, 9 and 12. Data will be obtained through remote review of wireless data transmitted from each device.
Adherence/Compliance with NIV | 1 year
  Average time used on days used. Measured at week 1-2, months 1, 3, 6, 9 and 12. Data will be obtained through remote review of wireless data transmitted from each device.
Adherence/Compliance with NIV | 1 year
  Average time used on all days. Measured at week 1-2, months 1, 3, 6, 9 and 12. Data will be obtained through remote review of wireless data transmitted from each device.
Sleep assessed by type 3 portable monitors and transcutaneous capnography | 1 year
  At baseline
Epworth Sleepiness Scale assessment for daytime sleepiness | 1 year
  8 question survey that measures the propensity of falling asleep in different situations. Composite score reported, with a range from 0-24, the higher the score indicating a greater propensity for falling asleep. Administered at baseline, 1, 3, 6, 9 and 12 months
Insomnia Severity Index assessment for difficulty falling asleep and staying asleep. | 1 year
  7-item survey that uses a likert scale. Measures the nature, severity, and impact of insomnia in adults. Composite score reported (0-28), with a higher score indicating a greater severity of insomnia. Administered at baseline, 1, 3, 6, 9 and 12 months
Pittsburgh sleep quality index (PSQI) questionnaire to measure sleep disturbance and sleep habits | 1 year
  19 item questionnaire with 7 domains (sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction), using a likert scale. Measures sleep disturbance and usual sleep habits during the prior month only. A global socre of 0-21 is used, with a score >5 indicating poor sleep quality. The higher the score the poorer the sleep quality. Administered at baseline, 1, 3, 6, 9 and 12 months
Functional Outcomes of Sleep Questionnaire (short form) to measure functional status resulting from sleepiness and is a measure of sleep-related HRQoL. | 1 year
  10 item questionnaire with 5 subscales. Subscale scores are averaged to obtain a total score ranging from 5-20, with a higher score indicating better functional status. Administered at baseline, 1, 3, 6, 9 and 12 months
Utilization of healthcare services (visits to outpatient clinics and emergency services, and number of inpatient admissions) | 1 year
  Visits (both outpatient and inpatient) will be identified based on VA-specific stop codes which define what type of visit occurred (specialty, date, and provider type).

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Sarmiento, MD, MPH, Principal Investigator — San Francisco VA Health Care System
Locations (1):
- San Francisco VA Health Care System, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murphy PB, Rehal S, Arbane G, Bourke S, Calverley PMA, Crook AM, Dowson L, Duffy N, Gibson GJ, Hughes PD, Hurst JR, Lewis KE, Mukherjee R, Nickol A, Oscroft N, Patout M, Pepperell J, Smith I, Stradling JR, Wedzicha JA, Polkey MI, Elliott MW, Hart N. Effect of Home Noninvasive Ventilation With Oxygen Therapy vs Oxygen Therapy Alone on Hospital Readmission or Death After an Acute COPD Exacerbation: A Randomized Clinical Trial. JAMA. 2017 Jun 6;317(21):2177-2186. doi: 10.1001/jama.2017.4451. PMID 28528348
- [Background] Budweiser S, Hitzl AP, Jorres RA, Heinemann F, Arzt M, Schroll S, Pfeifer M. Impact of noninvasive home ventilation on long-term survival in chronic hypercapnic COPD: a prospective observational study. Int J Clin Pract. 2007 Sep;61(9):1516-22. doi: 10.1111/j.1742-1241.2007.01427.x. PMID 17686094
- [Background] De Backer L, Vos W, Dieriks B, Daems D, Verhulst S, Vinchurkar S, Ides K, De Backer J, Germonpre P, De Backer W. The effects of long-term noninvasive ventilation in hypercapnic COPD patients: a randomized controlled pilot study. Int J Chron Obstruct Pulmon Dis. 2011;6:615-24. doi: 10.2147/COPD.S22823. Epub 2011 Nov 18. PMID 22135493
- [Background] Storre JH, Matrosovich E, Ekkernkamp E, Walker DJ, Schmoor C, Dreher M, Windisch W. Home mechanical ventilation for COPD: high-intensity versus target volume noninvasive ventilation. Respir Care. 2014 Sep;59(9):1389-97. doi: 10.4187/respcare.02941. Epub 2014 Jul 29. PMID 25074944
- [Background] Oscroft NS, Chadwick R, Davies MG, Quinnell TG, Smith IE. Volume assured versus pressure preset non-invasive ventilation for compensated ventilatory failure in COPD. Respir Med. 2014 Oct;108(10):1508-15. doi: 10.1016/j.rmed.2014.07.010. Epub 2014 Jul 23. PMID 25123526
- [Background] Mansfield D, Naughton MT. Effects of continuous positive airway pressure on lung function in patients with chronic obstructive pulmonary disease and sleep disordered breathing. Respirology. 1999 Dec;4(4):365-70. doi: 10.1046/j.1440-1843.1999.00206.x. PMID 10612570
- [Background] Gunduz C, Basoglu OK, Tasbakan MS. Prevalence of overlap syndrome in chronic obstructive pulmonary disease patients without sleep apnea symptoms. Clin Respir J. 2018 Jan;12(1):105-112. doi: 10.1111/crj.12493. Epub 2016 Jun 6. PMID 27148977